CLINICAL TRIAL: NCT05720663
Title: Predicting Outcomes in Nonalcoholic Steatohepatitis With Advanced Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20024296; 1R01DK129564 (NIH)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nonalcoholic steatohepatitis (NASH): Adult patients nonalcoholic steatohepatitis (NASH)
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Participants will receive the standard of care for their condition

SUMMARY:
Nonalcoholic Steatohepatitis (NASH) is a condition with increased amount of fat, inflammation and scarring in the liver. In compensated cirrhosis, the liver is coping with this damage and maintaining its important functions. Decompensation occurs when the liver becomes unable to perform all of its functions adequately. Variceal hemorrhage (bleeding from abnormal vessels in the liver called varices), Ascites (abnormal build-up of fluid in the abdomen), and Encephalopathy (brain confusion as a result of the liver not being able to get rid of toxic substances) are three symptoms of liver decompensation.

The purpose of this research study is to investigate better ways to routinely monitor the condition of patients with NASH with compensated cirrhosis and to better pinpoint the development of decompensation in the livers of these patients.

DETAILED DESCRIPTION:
This clinical research study is done to investigate better ways to routinely monitor the condition of patients with Nonalcoholic Steatohepatitis (NASH) with compensated cirrhosis. The purpose of this study is to better pinpoint the development of decompensation in the livers of these patients (some symptoms are variceal hemorrhage, ascites, and encephalopathy, defined below).

NASH is a condition with increased amount of fat, inflammation and scarring in the liver. In compensated cirrhosis, the liver is coping with this damage and maintaining its important functions. Decompensation occurs when the liver becomes unable to perform all of its functions adequately. Variceal hemorrhage (bleeding from abnormal vessels in the liver called varices), Ascites (abnormal build-up of fluid in the abdomen), and Encephalopathy (brain confusion as a result of the liver not being able to get rid of toxic substances) are three symptoms of liver decompensation.

Aside from current routine procedures including blood draws, this study will check to see how effectively adding three additional procedures will help predict development of liver decompensation. These additional procedures are Spleen Stiffness Measurement (SSM) during a special liver ultrasound called a Fibroscan, an imagining scan called Magnetic Resonance Imagining (MRI) using a contrast agent called Gadoxetate Sodium to highlight cirrhosis, and an MRI scan called metabophenotype, which examines muscle composition of the liver.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with presence of NAFLD associated cirrhosis.

* Cirrhosis: biopsy confirmed or Agile F (F4) score > 0.45
* NAFLD as an etiology of liver disease will be determined based on presence of any of the following:

  * Biopsy showing >5% steatosis or
  * CAP > 280 dB/m or MR-PDFF>5%
  * If CAP < 280 dB/m or MR-PDFF <5%, then must have type 2 diabetes and or 2 or more features of metabolic syndrome for 5 years (cryptogenic cirrhosis)

Exclusion Criteria:

* Refusal to consent
* Alcohol use > 14/21 gm/week cutoff
* Other causes of chronic liver disease
* MELD > 12
* Hepatic and extrahepatic cancers expected to limit life expectancy < 2 yrs
* prior hepatic resections, TIPS, splenic embolization
* prior decompensation events
* inability to fit into MRI (failed hula-hoop test)
* general contraindication for MRI contrast (GFR < 30 ml/min)
* contraindications for MRI
* pregnancy
* acute kidney injury
* reduced kidney function (GFR <30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with presence of NAFLD associated cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of deaths | Up to 2 years
  Number of deaths will be determined from death records and patient charts.
Incidents of variceal hemorrhage | Up to 2 years
  Number of participants showing bleeding from abnormal vessels in the liver called varices will be assessed using an endoscopy exam.
Incidents of ascites | Up to 2 years
  Number of participants with experiencing abnormal build-up of fluid in the abdomen will be assessed using a clinical exam including an ultrasound graded per clinical standards.
Hepatic Encephalopathy (HE) | Up to 2 years
  Number of grade 2, 3, or 4 HE events will be assessed by clinician during exams.

SECONDARY OUTCOMES:
Model For End-Stage Liver Disease (MELD) score | Up to 2 years
  Number of participants with MELD scores greater than 15
Hepatocellular cancer (HCC) | Up to 2 years
  Number of participants with HCC

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Siddiqui, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No